CLINICAL TRIAL: NCT00009581
Title: Targeted Delivery of Nitric Oxide by Hemoglobin to Improve Regional Blood Flow in Sickle Cell Disease
Brief Title: Nitric Oxide to Improve Blood Flow in Sickle Cell Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010078; 01-CC-0078
Record Dates: First submitted 2001-02-01; First posted 2001-02-02 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-01

CONDITIONS: Sickle Cell Anemia
Keywords: Endothelial Function; Hydroxyurea; Leukocyte Gene Expression; Nitrosylated Hemoglobin; Sickle Cell Anemia; Nitric Oxide
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — omega-N-Methylarginine; Acetylcholine

INTERVENTIONS:
Drug: L-NMMA
Drug: Acetylcholine

SUMMARY:
Nitric oxide is important in regulating blood vessel dilation, and consequently, blood flow. This gas is continuously produced by cells that line the blood vessels. It is also transported from the lungs by hemoglobin in red blood cells. This study will examine how this gas regulates blood vessels and blood flow in people with sickle cell anemia. It will also look at a possible benefit of using certain genetic information to compare the white blood cells of people with sickle cell anemia to those without the disease.

Patients with sickle cell anemia and healthy normal volunteers 18 to 65 years of age may be eligible for this study. Candidates will be screened with a medical history, cardiovascular physical examination, electrocardiogram and routine blood tests. Participation of volunteers without sickle cell anemia will be limited to a single blood draw for genetic study. Sickle cell disease patients will undergo the following procedures:

Patients will lie in a reclining chair during the study. After administration of a local anesthetic, small tubes will be inserted through a needle into the artery and vein of the patient's forearm. These are used to measure blood pressure and draw blood samples during the study. Forearm blood flow will be measured using pressure cuffs placed on the wrist and upper arm, and a strain gauge (a rubber band device) placed around the forearm. When the cuffs are inflated, blood flows into the arm, stretching the strain gauge, and the flow measurement is recorded. A small lamp will be positioned over the hand. Light reflected back from the hand provides information about nitric oxide and hemoglobin in the blood of the skin. A squeezing device called a dynamometer will be used to measure handgrip strength.

Baseline blood flow, nitric oxide, hemoglobin, and handgrip will be measured after an infusion of glucose (sugar) and water. These measurements will be repeated at various times before, during and after administration of small doses of the following drugs:

* Sodium nitroprusside - causes blood vessels to dilate and increases blood flow to the heart
* Acetylcholine - causes blood vessels to dilate and slows heart rate
* LNMMA - decreases blood flow by blocking the production of nitric oxide

There will be a 20- to 30-minute rest period between injections of the different drugs.

When the above tests are completed, the patient will breathe a mixture of room air and nitric oxide for 1 hour through a facemask placed over the face, after which forearm blood flow and light reflected from the hand will be measured. Then the patient will do the handgrip exercise for 5 minutes, after which blood flow and hand lamp measurements will be taken. After a 20-minute rest period (with continued breathing of room air/nitric oxide), L-NMMA will be infused again. The handgrip exercise, blood flow and hand lamp measurements will be repeated. The face mask will then be removed, and the tubes will be removed 20 minutes later.

Blood samples will be collected at various times during the 5- to 6-hour study through the tubes in the arm. Some of the blood will be used to look at genes that make proteins involved in cell-to-cell communication, inflammation, and in making red and white blood cells stick to the lining of blood vessels.

DETAILED DESCRIPTION:
Sickle cell anemia is an autosomal recessive disorder and the most common genetic disease affecting African-Americans. Approximately 0.15% of African-Americans are homozygous for sickle cell disease, and 8% have sickle cell trait. Acute pain crisis and acute chest syndrome are common complications of sickle cell anemia. Inhaled nitric oxide (NO) has been proposed as a possible therapy for the acute chest syndrome. Anecdotally, NO has been described to rapidly improve the hypoxemia and the clinical course of the acute chest syndrome. Furthermore, a number of recent studies have suggested that NO may have a favorable impact on sickle red cells at the molecular level and could improve the abnormal microvascular perfusion that is characteristic of sickle cell anemia. This clinical trial is designed to test the hypotheses that 1) individuals with sickle cell anemia have endothelial dysfunction with reduced local synthesis and release of NO, that may reduce regional perfusion at rest and impair the vasodilator response to stress, and 2) during NO inhalation, delivery of NO bound to hemoglobin will be enhanced and will improve these abnormalities in regional vascular perfusion. Studies will be performed on untreated sickle cell anemia patients and on patients managed with chronic hydroxyurea therapy. Demonstration of improved regional perfusion with NO therapy could have significant implications for patient management during acute pain crisis and the acute chest syndrome.

ELIGIBILITY:
INCLUSION CRITERIA

Males or females 18 to 65 years of age are eligible.

Diagnosis of sickle cell disease (electrophoretic documentation of SS, SC, or S beta(0) thallassemia genotype is required).

Hematocrit greater than 18 percent (with an absolute reticulocyte count greater than 100,000/ml).

Volunteer subjects taking hydroxyurea must have been on therapy with the drug for at least four months. Volunteer subjects not taking hydroxyurea must have been off of therapy with the drug for at least 4 months.

EXCLUSION CRITERIA

Clinically unstable sickle cell anemia defined as having an acute pain crisis within the last week.

Age less than 18 years or greater than 65 years.

Current pregnancy or lactation.

Conditions that may independently affect endothelial function:

1. Diabetes mellitus or Fasting blood sugar greater than 120 mg/dL
2. Cigarette smoking within two years
3. Hypertension (diastolic blood pressure greater than 90 mmHg)
4. Lipid abnormalities (LDL cholesterol greater than 160 mg/dL, HDL cholesterol less than 30 mg/dL, triglycerides greater than 500 mg/dL)
5. Creatinine greater than 1.0 mg/dL

Hematocrit less than or equal to 18 percent: however, patients may return for evaluation at a later date.

No aspirin or non-steroidal antiinflammatory drugs (NSAIDs for one week and caffeine the day of the study). Patients on opiates and acetaminophen will not be excluded.

Patients taking sildenafil (Viagra) will be excluded from the study.

Recent transfusion (last 4 weeks) or hemoglobin A greater than 5 percent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 65
Dates: Start 2001-01; Study Completion 2003-01

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Atz AM, Wessel DL. Inhaled nitric oxide in sickle cell disease with acute chest syndrome. Anesthesiology. 1997 Oct;87(4):988-90. doi: 10.1097/00000542-199710000-00037. No abstract available. PMID 9357905
- [Background] Belcher JD, Marker PH, Weber JP, Hebbel RP, Vercellotti GM. Activated monocytes in sickle cell disease: potential role in the activation of vascular endothelium and vaso-occlusion. Blood. 2000 Oct 1;96(7):2451-9. PMID 11001897
- [Background] Cardillo C, Kilcoyne CM, Cannon RO 3rd, Panza JA. Racial differences in nitric oxide-mediated vasodilator response to mental stress in the forearm circulation. Hypertension. 1998 Jun;31(6):1235-9. doi: 10.1161/01.hyp.31.6.1235. PMID 9622135